CLINICAL TRIAL: NCT07246304
Title: A Preliminary Exploratory Clinical Study of TC-D101 in the Treatment of DLL3-Positive Relapsed/Refractory Primary Small Cell Lung Cancer
Brief Title: TC-D101 Cell Therapy for Patients With DLL3-Positive SCLC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: TCRCure Biopharma Ltd. (Industry)
Collaborators: The Jinling Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D101-IIT-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Small Cell Lung Cancer ( SCLC ); CAR-T Cell Therapy
Keywords: Small Cell Lung Cancer ( SCLC ); CAR-T Cell Therapy; DLL3
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TC-D101 CAR-T Cell Therapy (Experimental): Following lymphodepletion chemotherapy, participants will receive Following lymphodepletion chemotherapy, participants will receive TC-D101 CAR-T Cell CAR-T
  Interventions: Biological: TC-D101 CAR-T

INTERVENTIONS:
Biological: TC-D101 CAR-T — TC-D101 CAR-T treatment follows a lymphodepletion Drug: Fludarabine and Cyclophosphamide.
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
This is a single-arm, open-label, dose-escalation clinical trial designed to evaluate the safety, tolerability, expansion, and persistence of TC-D101 CAR-T cells in patients with DLL3-positive Relapsed/Refractory primary small cell lung cancer(r/r SCLC) who have progressed after prior therapies. The primary objective is to determine the maximum tolerated dose (MTD), with a secondary aim to assess preliminary clinical efficacy in SCLC.

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label, single-dose clinical trial to evaluate the safety and efficacy of TC-D101 CAR-T cell therapy in patients with r/r SCLC. The study protocol consists of five main stages: (1) patient screening, (2) collection of peripheral blood mononuclear cells (PBMCs), (3) lymphodepletion chemotherapy, (4) TC-D101 CAR-T cell infusion, and (5) post-infusion follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily provide written informed consent.
2. Aged 18-75 years (inclusive).
3. Life expectancy ≥ 3 months.
4. ECOG performance status 0-1.
5. Failed or unsuitable for standard therapy.
6. At least one measurable lesion per RECIST 1.1.
7. DLL3-positive r/r SCLC confirmed by immunohistochemistry.
8. Adequate organ and bone marrow function.
9. Effective contraception required for participants of childbearing potential.
10. Adequate venous access for leukapheresis.

Exclusion Criteria:

1. Primary CNS malignancy or uncontrolled CNS metastases.
2. Other malignancies within 5 years (except adequately treated non-melanoma skin cancer or carcinoma in situ).
3. Active autoimmune disease or history of autoimmune disease.
4. Immunodeficiency, including HIV positivity.
5. Bleeding disorders (inherited or acquired).
6. Clinically significant cardiovascular disease.
7. Active infection (including tuberculosis, hepatitis B/C, syphilis).
8. Pregnant or breastfeeding women.
9. Clinically significant ascites . 10 Uncontrolled pleural effusion or pericardial effusion.

11. Prior cell or gene therapy. 12. Severe drug hypersensitivity history. 13. Investigator-assessed unsuitability for trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of TC-D101 CAR-T cells | Up to 24 months
  The incidence, type, and severity of all adverse events, serious adverse events, and abnormal laboratory findings.
Safety of TC-D101 CAR-T cells | Up to 1 month
  Incidence of DLT

SECONDARY OUTCOMES:
Efficacy of TC-D101 CAR-T cells | Up to 24 months
  Optimal objective response rate (ORR)

OTHER OUTCOMES:
To investigate the Cmax of TC-D101 CAR-T cells in the peripheral blood after infusion | Up to 24 months
To assess TC-D101 CAR-T cell trafficking into tumor tissues after infusion | Up to 24 months
  To detect TC-D101 CAR-T cell number in tumor tissues after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- The Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No